CLINICAL TRIAL: NCT01533675
Title: A Comparison Study of the Tensile Strength of Sutures Used in Dermatologic Surgery on the Day of Suture Removal, Following Wound Care With Two Different
Brief Title: A Comparison Study of the Tensile Strength of Sutures Used in Dermatologic Surgery on the Day of Suture Removal, Following Wound Care With Two Different Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Keyvan Nouri, M.D Professor of Dermatology, Ophthalmology & Otolaryngology, Chief of Dermatology Servic, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # 20100301
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Sutured Wounds
Keywords: suture, tensile strength, wound care, saline, hydrogen peroxide, skin closure, wounds, wound healing, wound cleansing, antiseptics
MeSH Terms: conditions — Wounds and Injuries | interventions — Hydrogen Peroxide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrogen peroxide (Experimental)
  Interventions: Other: Hydrogen peroxide
- Saline (Active Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Hydrogen peroxide — Once daily topical application of 3% hydrogen peroxide using a cotton-tipped applicator
  Arms: Hydrogen peroxide
Other: Saline — Once daily topical application of normal saline, using a cotton-tipped applicator
  Arms: Saline

SUMMARY:
Sutures are an integral part of surgery and available materials are diverse, as are the options for post-procedure care. Both saline and hydrogen peroxide are commonly used cleansing agents. This study aims to compare the effect of saline and hydrogen peroxide on the tensile strength of 4-0 nylon sutures following removal from a cutaneous surgical wound.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to comply with the informed consent procedures
* Subject's wound is on the body or scalp
* Subject will be able to come to the clinic for suture removal on day 14

Exclusion Criteria:

* Subject is less than 18 years of age
* Subject's wound was not closed with 4-0 nylon sutures
* Subject's wound is on the face
* Subject plans to apply other topicals to the area under study
* Subject's suture is removed before or after day 14

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Tensile strength of 4-0 nylon sutures | 14 days
  The tensile strength was defined as the force required to break the suture, with breaking strength as the maximum strength that a material can withstand when subjected to an applied load, without taking into consideration the cross sectional area. The strength of the sutures was measured using a tensometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Result] Snyder CC. On the history of the suture. Plast Reconstr Surg. 1976 Oct;58(4):401-6. doi: 10.1097/00006534-197610000-00001. No abstract available. PMID 785506
- [Result] Hochberg J, Meyer KM, Marion MD. Suture choice and other methods of skin closure. Surg Clin North Am. 2009 Jun;89(3):627-41. doi: 10.1016/j.suc.2009.03.001. PMID 19465201